CLINICAL TRIAL: NCT06637137
Title: Patient Blood Management in Cardiac Surgical Patients: the ICARUS-2 Study
Brief Title: Patient Blood Management in Patients Scheduled for Cardiac Surgery
Acronym: ICARUS-2
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, CORSI FILIPPO, Meidcal doctor, principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6727/2024; FPG gemelli IRCCS (Other: FPG gemelli IRCCS)
Record Dates: First submitted 2024-10-06; First posted 2024-10-15 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Anemia; Anemia, Iron-Deficiency; Iron Deficiency Anemia Treatment; Iron Deficiency Anemia (IDA); Cardiac Surgical Patients; Blood Loss, Surgical
Keywords: iron; anemia; cardiac surgery; patient blood management
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Blood Loss, Surgical | interventions — Iron; Folic Acid; Vitamin B Complex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Prospectic cohort: patients scheduled for cardiac surgery who fulfil the inclusion criteria
  Interventions: Drug: Iron
- retrospective cohort ICARUS 1: patients scheduled for cardiac surgery (2021) with a known iron status, treated if indicated 1 or 2 days before surgery with iron supplementation.
- retrospective cohort: patients scheduled for cardiac surgery (2019-2020)with an unknown iron status and never treated with iron supplementation

INTERVENTIONS:
Drug: Iron — Patients who present a state of hypoferritinemia or a state of reduced transferrin saturation will undergo administration of i.v iron at least 2 weeks before scheduled cardiac surgery, plus acid folic and B vitamin co-administration.
  Other Names: folic acid; b vitamin
  Groups: Prospectic cohort

SUMMARY:
The ICARUS 2 study has the general objective of collecting data in patients undergoing cardiac surgery; in our centre, in order to optimize and improve hemoglobin values, a team of haematologists, assisted by cardio anesthetists and cardiac surgeons, will evaluate the blood tests of patients scheduled for elective cardiac surgery in order to correct any states of hypoferritinemia (low iron in the blood) to promote recovery from blood losses related to cardiac surgery. This objective is strongly encouraged by the good use of blood programs currently in force at our foundation.

In particular, the research presented here intends to demonstrate a reduction in the number of intra- and post-operative transfusions.

DETAILED DESCRIPTION:
A significant percentage of patients schduled for cardiac surgery have an absolute or relative iron deficiency (ID) with or without anemia. Preoperative outpatient treatment of anemia and iron deficiency is one of the pillars of patient blood management (PBM). Data collected at our institution show that 35% of patients undergoing cardiac surgery at the Foundation receive 2 or more units of concentrated red blood cells at surgery or in the following 7 days. A recently published ambispective study (ICARUS) demonstrated that intravenous iron supplementation, even in the immediate pre-operative period (i.e 1 or 2 days), reduces the number of post-operative transfusions and the length of hospital stay. Similar results were recently obtained by other authors in a randomized study. Assuming the correction of ID at an earlier stage, the haematological outcome could be significantly better, with a reduction in the percentage of patients transfused and in the average transfusion requirement, increase in haemoglobin levels at discharge, improvement in clinical conditions and possible further reduction of the length of stay. All this could translate into a further reduction in costs related to the intervention.

The study is observational and involves the early application of the PBM program based on good clinical practice which includes the correction of absolute or relative ID. This deficiency will be treated at least 2 weeks before the planned cardiac surgery: the patient will receive an i.v. of iron in the clinic, in accordance with the indications, doses and route of administration for which the use of the drug is approved and the drug distributed on the market. At the same time as iron administration, vitamin supplementation will be prescribed (Vitamin B12 1 mg total subcutaneously) and oral folic acid (5 mg/day).

ELIGIBILITY:
Inclusion Criteria:

- all adult patients scheduled for elective cardiac surgery

Exclusion Criteria:

* pregnancy
* dyalisis
* patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients candidate for elective cardiac surgery at our tertiary care hospital are eligible for the study purpose.
Sampling Method: Probability Sample
Enrollment: 464 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients receiving RBC transfusion within post-operative day 7 | within post operative day 7
  number of RBC units transfused from the operating room till post operative day 7

SECONDARY OUTCOMES:
cost measured in euros for the IDA treatment and blood product consumption | from enrollment to 1 week after surgery
  We will assess if ID screening and iron replacement is cost-effective, considering the costs, expressed in euros, of the treatment with ferric carboxymaltose, folic acid and B12 vitamin, the pRBC consumption and hospitalization (either in ICU or in the regular ward).
Hb values at last postoperative control within 7 days from surgery | within post operative day 7
  Hb values at last postoperative control within 7 days from surgery
ICU lenght of stay | through study completion, an average of 2 year
  lenght of stay in ICU
Number of allogenic blood products administered | within the first 7 days post operative
  Number of allogenic blood products administered (i.e fresh frozen plasma or platelet units).
mortality | from surgery within post operative day 7
  patients died within the first 7 days after surgery
Hospital Lenght of Stay | through study completion, an average of 2 year
  The number of days spent in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: luciana Teofili, Phd, Study Director — Fondazione Policlinico Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
IPPD will be shared upon reasonable request to the PPI and after approval of ethic commitee.

REFERENCES:
- [Background] Corsi F, Pasquini A, Guerrera M, Bevilacqua F, Taccheri T, Antoniucci ME, Calabrese M, Valentini CG, Orlando N, Bartolo M, Cannetti G, Pellegrino C, Cavaliere F, Teofili L. Single shot of intravenous iron in cardiac surgery: The ICARUS study. J Clin Anesth. 2023 Feb;84:111009. doi: 10.1016/j.jclinane.2022.111009. Epub 2022 Nov 16. PMID 36401886
- See also: Intravenous iron administration before cardiac surgery reduces red blood cell transfusion in patients without anaemia. — https://pubmed.ncbi.nlm.nih.gov/37838604/
- See also: Effect of ultra-short-term treatment of patients with iron deficiency or anaemia undergoing cardiac surgery: a prospective randomised trial. — https://pubmed.ncbi.nlm.nih.gov/31036337/
- See also: Iron supplementation for patients undergoing cardiac surgery: a systematic review and meta-analysis of randomized controlled trials. — https://pubmed.ncbi.nlm.nih.gov/34559371/